CLINICAL TRIAL: NCT02565043
Title: A Prospective, Open, Multi-centre Study to Evaluate Clinical Efficacy, Functionality and Device Performance of a New Portable Negative Pressure Wound Therapy System (RENASYS TOUCH) in the Management of Acute, Sub-acute and Chronic Wounds
Brief Title: The Clinical Efficacy of RENASYS TOUCH NPWT System in the Management of Acute, Sub-acute and Chronic Wounds
Acronym: NPWT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT13/01
Record Dates: First submitted 2015-09-28; First posted 2015-10-01 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Wound and Injuries; Surgical Wound Dehiscence
Keywords: Negative Pressure Wound Therapy
MeSH Terms: conditions — Wounds and Injuries; Surgical Wound Dehiscence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RENASYS TOUCH Negative Pressure Wound Therapy Device (Experimental): Active Device: "RENASYS TOUCH NPWT" device administered to all patients using the intermittent/variable therapy mode, for up to 28 days of therapy.
  Interventions: Device: RENASYS TOUCH Negative Pressure Wound Therapy System
- RENASYS TOUCH Negative Pressure Wound Therapy System (Active Comparator): Active Device: "RENASYS TOUCH NPWT" device administered to all patients using the continuous therapy mode for up to 28 days of therapy.
  Interventions: Device: RENASYS TOUCH Negative Pressure Wound Therapy System

INTERVENTIONS:
Device: RENASYS TOUCH Negative Pressure Wound Therapy System — RENASYS TOUCH NPWT System was administered to all participants.
  Other Names: "RENASYS TOUCH NPWT" System

SUMMARY:
The study is looking at the clinical efficacy, functionality and device performance of a new Negative Pressure Wound Therapy (NPWT) system in the management of a variety of wound types, in a real-life clinical setting. The study will comprise a prospective, open-labeled, multi-center study in a number of care-settings (both hospital and community) in South Africa. The patient's reference wound will be randomized to treatment with either intermittent or continuous NPWT mode to assess whether the delivery of NPWT via each of these therapy settings will have an effect on the rate and quality of wound healing.

DETAILED DESCRIPTION:
The study will comprise a prospective, open-labeled, multi-center study to assess the clinical efficacy, functionality and device performance of the new portable negative pressure wound therapy system in the management of acute, sub-acute and chronic wounds.

The patient's reference wound will be randomized to treatment with either intermittent or continuous NPWT mode to ensure minimum numbers in each group for analysis.

The primary objective of the study is to determine the time (days) to achieve the point where the reference wound is ready to be closed either by surgical intervention (STSG, simple flap or suturing) or by secondary intention.

ELIGIBILITY:
Inclusion Criteria:

* The patient is able to understand the study and is willing to consent to the study
* The patient consents to the on-going use of their de-identified photos by the Sponsor for purposes outside of this study
* Patients must be at least 18 years old
* Males and females. If female, they must not be pregnant. If female and of reproductive age, a pregnancy test will be provided
* Patient must have an acute, sub-acute or chronic wound that would benefit from the application of topical Negative Pressure Wound Therapy (NPWT)
* Patients must have an acute or sub-acute wound requiring wound bed preparation for an expected minimum of 4 days in advance of either planned surgical closure (including delayed primary closure, flaps or grafts) or planned secondary closure, OR a chronic wound requiring wound bed preparation in advance of planned surgical closure (not secondary intention)
* The patient, or the patient's legal representative, if the patient is incapable of giving legal consent, is able to understand the trial and is willing to consent to the trial

Exclusion Criteria:

* Patients with a known history of poor compliance with medical treatment.
* Patients who have participated in this study previously and who [healed or] were withdrawn.
* Patients who are unable to understand the aims and objectives of the study.
* Presence of necrotic tissue, or >25% slough in the reference wound bed. Once debridement has taken place, treatment with the investigational product may proceed
* Patients whose reference wound displays evidence of extensive tunnelling or sinus tracts
* Previously confirmed and untreated osteomyelitis
* Malignancy in the reference wound
* Non-enteric and unexplored Fistulas
* Presence of untreated infection in the reference wound bed (Infection must be treated with systemic antibiotics to permit inclusion in the trial and can be administered concurrently during the trial treatment regime)
* Active bleeding. Once haemostasis has been achieved, treatment with the investigational product may proceed
* Exposure of blood vessels or organs at the base of the reference wound
* Patients with a known history of poor compliance with medical treatment
* Patients who have participated in this trial previously and who healed or were withdrawn
* Patients treated on an out-patient basis who cannot continue to be treated as out-patients and/or attend the clinic for dressing changes as detailed in the treatment regimen of the study protocol
* Patients whose wounds are not suitable for treatment with intermittent therapy mode (e.g. highly exuding wounds, wounds with tunnels or undermining, wounds in difficult areas where maintaining a seal is problematic, patients who experience severe pain during intermittent therapy)
* Patients who are employees of Smith & Nephew group companies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-04; Primary Completion 2016-08 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
The time to achieve the point where the reference wound is ready to be closed either by surgical intervention (STSG, simple flap or suturing) or by secondary intention | 28 days

SECONDARY OUTCOMES:
To determine the percentage of wounds that are ready to be closed either by surgical intervention (STSG, simple flap or suturing) or by secondary intention | 28 days
To assess the percentage of wounds that are ready to be closed either by surgical intervention (STSG, simple flap or suturing) or by secondary intention, in wounds that are randomized to intermittent or continuous therapy mode | 28 days
The percentage change in wound area | 28 days
  To assess progress towards wound closure using the percentage change in wound area (cm2)
The number of patients with a confirmed clinical infection or presenting with clinical signs of infection | 28 days
  Patients that have a confirmed clinical infection or the number of patients that present with clinical signs of infection in their reference wound
The number of patients with the condition of their surrounding skin recorded as either Healthy, Fragile, Inflamed, Macerated, Dry and Flaky, or Other | 28 days
  To assess the condition of the patients surrounding skin
To record the patients level of pain using a 10-point pain scale, on application and during therapy, in patient's wounds that are randomised to intermittent or continuous therapy mode | 28 days
  To assess the patients level of pain on application and during therapy
The study will monitor safety in use and will record and assess all adverse events that occur during the study | 28 days
The percentage change in wound volume | 28 days
  To assess progress towards wound closure using the percentage change in wound area (cm3)
The percentage change in wound depth | 28 days
  To assess progress towards wound closure using the percentage change in wound depth (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Forlee, MD, Principal Investigator — Dr Matley & Partners
Locations (2):
- South Africa (2):
  - Tiervlei Trail Centre, Bellville, Cape Town
  - Dr Matley & Partners, Claremont, Cape Town

REFERENCES:
- [Background] Morykwas MJ, Argenta LC, Shelton-Brown EI, McGuirt W. Vacuum-assisted closure: a new method for wound control and treatment: animal studies and basic foundation. Ann Plast Surg. 1997 Jun;38(6):553-62. doi: 10.1097/00000637-199706000-00001. PMID 9188970
- [Background] Argenta LC, Morykwas MJ. Vacuum-assisted closure: a new method for wound control and treatment: clinical experience. Ann Plast Surg. 1997 Jun;38(6):563-76; discussion 577. PMID 9188971
- [Background] Krug E, Berg L, Lee C, Hudson D, Birke-Sorensen H, Depoorter M, Dunn R, Jeffery S, Duteille F, Bruhin A, Caravaggi C, Chariker M, Dowsett C, Ferreira F, Martinez JM, Grudzien G, Ichioka S, Ingemansson R, Malmsjo M, Rome P, Vig S, Runkel N, Martin R, Smith J; International Expert Panel on Negative Pressure Wound Therapy [NPWT-EP]. Evidence-based recommendations for the use of Negative Pressure Wound Therapy in traumatic wounds and reconstructive surgery: steps towards an international consensus. Injury. 2011 Feb;42 Suppl 1:S1-12. doi: 10.1016/S0020-1383(11)00041-6. PMID 21316515
- [Background] Birke-Sorensen H, Malmsjo M, Rome P, Hudson D, Krug E, Berg L, Bruhin A, Caravaggi C, Chariker M, Depoorter M, Dowsett C, Dunn R, Duteille F, Ferreira F, Francos Martinez JM, Grudzien G, Ichioka S, Ingemansson R, Jeffery S, Lee C, Vig S, Runkel N; International Expert Panel on Negative Pressure Wound Therapy [NPWT-EP]; Martin R, Smith J. Evidence-based recommendations for negative pressure wound therapy: treatment variables (pressure levels, wound filler and contact layer)--steps towards an international consensus. J Plast Reconstr Aesthet Surg. 2011 Sep;64 Suppl:S1-16. doi: 10.1016/j.bjps.2011.06.001. Epub 2011 Aug 24. PMID 21868296
- [Background] Vig S, Dowsett C, Berg L, Caravaggi C, Rome P, Birke-Sorensen H, Bruhin A, Chariker M, Depoorter M, Dunn R, Duteille F, Ferreira F, Martinez JM, Grudzien G, Hudson D, Ichioka S, Ingemansson R, Jeffery S, Krug E, Lee C, Malmsjo M, Runkel N; International Expert Panel on Negative Pressure Wound Therapy [NPWT-EP]; Martin R, Smith J. Evidence-based recommendations for the use of negative pressure wound therapy in chronic wounds: steps towards an international consensus. J Tissue Viability. 2011 Dec;20 Suppl 1:S1-18. doi: 10.1016/j.jtv.2011.07.002. Epub 2011 Nov 25. PMID 22119531
- [Background] Hudson DA, Adams KG, Van Huyssteen A, Martin R, Huddleston EM. Simplified negative pressure wound therapy: clinical evaluation of an ultraportable, no-canister system. Int Wound J. 2015 Apr;12(2):195-201. doi: 10.1111/iwj.12080. Epub 2013 May 7. PMID 23647737
- [Background] Clare MP, Fitzgibbons TC, McMullen ST, Stice RC, Hayes DF, Henkel L. Experience with the vacuum assisted closure negative pressure technique in the treatment of non-healing diabetic and dysvascular wounds. Foot Ankle Int. 2002 Oct;23(10):896-901. doi: 10.1177/107110070202301002. PMID 12398140
- [Background] Mendonca DA, Cosker T, Makwana NK. Vacuum-assisted closure to aid wound healing in foot and ankle surgery. Foot Ankle Int. 2005 Sep;26(9):761-6. doi: 10.1177/107110070502600915. PMID 16174508
- [Background] McCallon SK, Knight CA, Valiulus JP, Cunningham MW, McCulloch JM, Farinas LP. Vacuum-assisted closure versus saline-moistened gauze in the healing of postoperative diabetic foot wounds. Ostomy Wound Manage. 2000 Aug;46(8):28-32, 34. PMID 11189545